CLINICAL TRIAL: NCT03243357
Title: In Vivo Assessment of Endodontics Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Camilla Christian Gomes Moura, Adjunct Professor of Endodontics of Faculty of Dentistry of Federal University of Uberlandia, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 68089517.2.0000.5152
Record Dates: First submitted 2017-07-26; First posted 2017-08-09 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Apical Periodontitis
Keywords: Endodontics, molars, instrumentation, obturation, anatomy
MeSH Terms: conditions — Periapical Periodontitis; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TF Adaptive (First Apical Binding File) (Experimental): Endodontic treatment(teeth with periapical periodontitis&radiolucence).Local anesthesia (4%Articaine with1:100,000 epinephrine),isolation with rubber dam&standard access cavity preparation.Using 2.5 %sodium hypochlorite,canal negotiation,glide path,coronal flaring with Sx(ProTaper),determining working length&first apical binding file.Intervention: Root canal instrumentation:TF Adaptive system with enlargement of the root canal performed with up to 3 files larger than the diameter of the initial apical file. Irrigation2.5%NaOCl&EDTA (Ethylenediaminetetraacetic acid)under activation with ultrasound. Irrigation with saline solution and placement of medication based on calcium hydroxide. After 14 days, obturation: gutta-percha&epoxy resin sealer.
  Interventions: Procedure: TF Adaptive (First Apical Binding File)
- TF Adaptive (Control) (Other): In the control group,endodontic treatment (teeth with periapical periodontitis&radiolucence). Local anesthesia(4% Articaine with 1:100,000 epinephrine), isolation with rubber dam&standard access cavity preparation. Using 2.5 % sodium hypochlorite, canal negotiation, determining working length&glide path. Root canal instrumentation:TF Adaptive system according to the protocol recommended by the manufacturer.Irrigation 2.5% NaOCl & EDTA(Ethylenediaminetetraacetic acid)under activation with ultrasound. Irrigation with saline solution and placement of medication based on calcium hydroxide. After 14 days, the canals will be obturated with gutta-percha and epoxy resin sealer.
  Interventions: Procedure: TF Adaptive (Control)

INTERVENTIONS:
Procedure: TF Adaptive (First Apical Binding File) — Procedure: TF Adaptive System NiTi (Nickel titanium) Endo File System (SybronEndo) The root canal instrumentation will be performed by the TF Adaptive features Adaptive Motion (Elements Motor).
  Procedure: Instrumentation based on protocol of First Apical Binding File The enlargement of the root canal will be performed with three files larger than the diameter of the previously established initial apical file.
  Arms: TF Adaptive (First Apical Binding File)
Procedure: TF Adaptive (Control) — Procedure: TF Adaptive System NiTi (Nickel titanium)Endo File System The root canal instrumentation will be performed by the TF Adaptive features Adaptive Motion (Elements Motor).
  Procedure: Instrumentation based on manufacturer's protocol The enlargement of the root canal will be performed according to the manufacturer's directions.
  Other Names: TF Adaptive (Manufacturer's protocol)
  Arms: TF Adaptive (Control)

SUMMARY:
In view of the wide variety of mechanized endodontic instrumentation systems, the ideal would be that the choose of this system based on the anatomical characteristics of the canal and the biological precepts. In teeth with lesions, contaminated dentin should be removed. However, in many systems, the manufacturer's approach disregards the fact that in wider root canal, instruments used in the apical third small diameter (less than 0.40 mm) may not touch the walls at the final apical. Therefore, the establishment of the initial apical file (LAI), the first instrument that measures the resistance of the walls in working length, could be a criterion in the choice of which system to use, and how many files work within the root canals after LAI determination. However, there is a lack of studies that demonstrate that LAI determination affects the degree of cleaning achieved, as well as the impact that LAI-based instrumentation may have on microcracks formation, canal transportation, postoperative pain and quality of obturation.In this way, the investigators propose a study in vivo performed, in patients from 8 to 18 years of age, therefore in large root canals. The protocol recommended by the manufacturer will be compared by means of a prospective randomized clinical trial, with the addition of the XP Endo finisher and with the protocol based on the initial apical file evaluating postoperative pain, exacerbation between the sessions, the quality of the obturation and periapical radiolucency repair. Considering that currently performing endodontic treatments using mechanized instruments is taught in undergraduate courses throughout the country, studies of this nature help the execution of a endodontics more critical and effective.

DETAILED DESCRIPTION:
Infected root canal treatments will be performed in two sessions with a TF Adaptive system (Protocol recommended by manufacturer (Group Control) vs. Protocol based on the initial apical file). The root canals will be completed after 14 days. Patients will record postoperative pain during the follow-up period (7 days) using a Visual analogue scale (VAS) and the change in periapical radiolucency will be assessed by periapical index (PAI) scores.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have in their mandibular or maxillary molar teeth apical periodontitis symptomatic or asymptomatic with apical radiolucence.

Exclusion Criteria:

* Patients with medical history compromises outcomes
* Atresic and root canals
* Root canals with curvature greater than 30 degrees
* Previously performed endodontics treatment.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-03-07 (Estimated); Study Completion 2020-11-03 (Estimated)

PRIMARY OUTCOMES:
Pain level | 7 days
  A Visual Analogue Scale VAS scale will be used for the postoperative pain level. The patients will noted their postoperative pain level according to the VAS scale during the follow-up period.

SECONDARY OUTCOMES:
Periapical radiolucence Repair | 6 and 12 months
  The change will be observed in periapical radiolucence in X-ray at the 6 and 12-month follow-up visit to assess the treatment outcome The outcome measure will be the change in periapical radiolucency as assessed by periapical index (PAI) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla C Gomes Moura, PhD, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil